CLINICAL TRIAL: NCT00867971
Title: Is Recombinant Growth Hormone Therapy Associated With Increased Intraoccular Pressure?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ilan Youngster, Assaf Harofeh Medical Center
Other Study IDs: 162/08
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-02

CONDITIONS: Growth Hormone Treatment; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- RGH treated
  Interventions: Other: Measuring intraoccular pressure
- Starting treatment with RGH
  Interventions: Other: Measuring intraoccular pressure

INTERVENTIONS:
Other: Measuring intraoccular pressure — Measurement of intraoccular pressure by tonometry

SUMMARY:
Recombinant growth hormone is a common therapy in the pediatric population. A number of associated side effects have been described. Several years ago, a case report was published concerning a child that was treated with RGH and developed acute glaucoma. To date no study has evaluated the connection.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years
* treatment with recombinant growth hormone

Exclusion Criteria:

* Underlying Chronic diseases
* Family history of eye diseases
* elevated occular pressure prior to starting treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children age 6-18 treated with growth hormone
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Intraoccular pressure in children treated with RGH | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf harofeh medical center, Ẕerifin, Israel

REFERENCES:
- [Derived] Youngster I, Rachmiel R, Pinhas-Hamiel O, Bistritzer T, Zuckerman-Levin N, de Vries L, Naugolny L, Eyal O, Braunstein R, Rachmiel M. Treatment with recombinant human growth hormone during childhood is associated with increased intraocular pressure. J Pediatr. 2012 Dec;161(6):1116-9. doi: 10.1016/j.jpeds.2012.05.024. Epub 2012 Jun 23. PMID 22727870